CLINICAL TRIAL: NCT01607996
Title: Phase 1 Study of Epidural Anesthesia on Pancreatic Perfusion and Clinical Outcome in Patients With Severe Acute Pancreatitis
Brief Title: Effect of Epidural Anesthesia on Pancreatic Perfusion and Clinical Outcome in Patients With Severe Acute Pancreatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Leo Buhler, Associate Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUG 02-0555
Record Dates: First submitted 2012-05-22; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Severe Acute Pancreatitis
Keywords: Epidural anesthesia; pancreatic perfusion; pancreatic necrosectomy
MeSH Terms: conditions — Pancreatitis | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient controlled intravenous analgesia (Active Comparator): Fentanyl (10 microg/ml) continuous intravenous infusion at a rate of 10 to 20 microg/h
  Interventions: Drug: Patient controlled intravenous analgesia
- Epidural anesthesia (Experimental): Carbostesin (0.1%) and Fentanyl (2 microg/ml) at a continuous flow of 6 to 15 ml/hour
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Epidural will be performed using carbostesin (0.1%), fentanyl (2 microg/ml) administered continuously at a rate of 6 to 15 ml/hour
  Arms: Epidural anesthesia
Drug: Patient controlled intravenous analgesia — Fentanyl 10 microg/ml at continuous flow of 10 to 20 microg/hour
  Arms: Patient controlled intravenous analgesia

SUMMARY:
The aim of the study is to evaluate the safety, the potential beneficial effect of epidural anesthesia on pancreatic perfusion and clinical outcome of patients with severe acute pancreatitis.

DETAILED DESCRIPTION:
High mortality in severe acute pancreatitis (AP) is linked to necrosis of the gland. Animal studies showed that epidural anesthesia (EA) restores pancreatic microcirculation and decreases the severity of AP. The aim of the study is to evaluate the safety of EA, its effect on pancreatic perfusion and clinical outcome of patients with AP.

ELIGIBILITY:
Inclusion Criteria:

* Acute pancreatitis with Ranson Criteria over 2, and/or CRP over 100, and or pancreatic necrosis on CT scan

Exclusion Criteria:

* Coagulation disorders
* Skin infection of the vertebral region

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-07; Primary Completion 2010-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events related to epidural anesthesia | Participants will be followed for the duration of hospital stay, an expected average of 2 to 5 weeks
  Adverse events related to epidural anesthesia include hypotensive episodes or infection of the catheter
Pancreatic perfusion measured by computerized tomography | On day 0 and day 2 or 3 after hospital admission

SECONDARY OUTCOMES:
Clinical outcome | Participants will be followed for the duration of hospital stay, an expected average of 2 to 5 weeks
  Lenght of stay, admission to intensive care unit, need for surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Demirag A, Pastor CM, Morel P, Jean-Christophe C, Sielenkamper AW, Guvener N, Mai G, Berney T, Frossard JL, Buhler LH. Epidural anaesthesia restores pancreatic microcirculation and decreases the severity of acute pancreatitis. World J Gastroenterol. 2006 Feb 14;12(6):915-20. doi: 10.3748/wjg.v12.i6.915. PMID 16521220